CLINICAL TRIAL: NCT00261430
Title: Schizophrenia Treatment Acceptance Response Trial: a 20-week, Open-label, Multicenter, Randomized Study Comparing the Effect of the "GAIN Acceptance Approach Verses the "Approach-as-usual" in Supporting Patient Acceptance of Long-acting Risperidone (Risperdal� CONSTA�) in Adults With Schizophrenia
Brief Title: A 2-year Study of Patients With Schizophrenia Who Are Treated With Long-acting Injectable Risperidone.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002893
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; acceptance; motivational enhancement therapy; long-acting risperidone; intramuscular injection; Treatment Guidebook; GAIN Acceptance Approach
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Behavioral: GAIN Acceptance Approach

SUMMARY:
The purpose of this study is to examine treatment practices of adult schizophrenia patients by their own doctors, and to assess patient outcomes when treated with long-acting risperidone injection over a two-year period of observation.

DETAILED DESCRIPTION:
Controlled clinical trials for treating schizophrenia often involve selected patients with common characteristics. It is recognized that schizophrenia are much more diverse than those in the clinical setting, and that physician's prescribing practices may vary. The objective of the study is to examine treatment practices for adult schizophrenic patients by their own physicians, and to assess patient outcomes when treated with long-acting risperidone injection. This is a 2-year, prospective, multi-center, longitudinal, observational study in adults with schizophrenia. Physicians will determine the appropriate treatment for their patients, according to their usual practice. Patients starting treatment with long-acting risperidone injections and meeting all the study criteria may enroll in the study. Patients will continue their treatment according to usual care by their physicians. Patients will be asked questions at baseline and every three months for a period of two years to assess: efficacy of the medication, how well the patient is functioning, use of healthcare resources (e.g., emergency room visits, hospitalizations) patient work status, quality of life and patient satisfaction with the medicine. Safety will be monitored throughout the study. A dose of 25, 37.5 or 50 mg of risperidone, administered every 2 weeks by intramuscular injection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* long-term use of antipsychotic medication and taking any oral antipsychotic for 4 weeks before the study
* stable with respect to disease symptoms and other medical conditions
* if female, using birth control.

Exclusion Criteria:

* At risk to self or others
* use of injectable antipsychotics within the past 6 months, of clozapine, or of investigational drugs within 30 days
* considered to be resistant to treatment
* pregnant or breast-feeding
* not using birth control.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
After 12 weeks of treatment, the percentage of patients accepting long-acting risperidone injection switched using the "Gain Acceptance Approach" compared with those switched using the "approach as usual"

SECONDARY OUTCOMES:
Clinical Global Impression of Severity (CGI-S) and Clinical Global Impression of Change (CGI-C) to measure disease severity; Patient Attitude/Satisfaction scale and Clinician Attitude/Satisfaction scale after 12 weeks of treatment, measuring satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP

REFERENCES:
- See also: Schizophrenia Treatment Acceptance Response Trial — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=347&filename=CR002893_CSR.pdf